CLINICAL TRIAL: NCT05617859
Title: A Multicenter, Open, One-arm Phase II Study of Ranvastinib Mesylate Capsules in the Treatment of Advanced Bone and Soft Tissue Sarcoma After Chemotherapy Failure
Brief Title: Lenvatinib for Advanced Bone and Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, associate chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZUSC-20
Record Dates: First submitted 2022-10-31; First posted 2022-11-16 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-02

CONDITIONS: Effectiveness; Sexuality
MeSH Terms: conditions — Sexuality | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib mesylate capsule (Other): Eligible subjects with bone and soft tissue sarcoma were selected and treated with the following treatment regimens:Subjects will receive Lenvatinib mesylate capsules, 8mg (body weight ≤60kg) or 12mg (body weight >60kg) orally once daily. Take the medicine about half an hour after meals (the time of taking the medicine should be the same as possible every day) and take it with warm water.
  Interventions: Drug: Lenvatinib mesylate capsule

INTERVENTIONS:
Drug: Lenvatinib mesylate capsule — Lenvatinib mesylate capsule, 8mg (body weight ≤60kg) or 12mg (body weight >60kg), orally, once daily. Take the medicine about half an hour after meals (the time of taking the medicine should be the same as possible every day) and take it with warm water.

SUMMARY:
A total of 60 patients with metastatic/surgically unresectable bone and soft tissue sarcomas who had previously received multi-target TKI therapy and failed were enrolled to evaluate the efficacy and safety.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of lenvatinib mesylate capsule in patients with metastatic/surgically unresectable bone and soft tissue sarcomas who had previously received multitarget TKI therapy and failed.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 10-70, both male and female.
2. The Eastern Collaborative Oncology Group (ECOG) physical status score was 0-1. Subjects with amputation can be relaxed up to 2 points.
3. The expected survival time was ≥3 months.
4. Subjects with bone and soft tissue sarcomas with distant metastases or locally advanced disease who were not considered suitable for surgical treatment by the investigator.
5. Patients who had been treated with apatinib or anlotinib in the past, and the efficacy was evaluated as CR\PR\SD\PD, and had no response to other systemic therapy after drug resistance, or had reprogression after more than 3 months.
6. There were measurable lesions that met RECIST1.1 criteria.
7. All acute toxicities from previous antitumor therapy or surgery resolved to grade 0-1 (according to NCI-CTCAE, version 4.03) or to enrollment/exclusion criteria by day 1 of the first cycle (C1D1), except for toxicities such as hair loss that the investigator considered to pose no safety risk to the subject.
8. Adequate organ and bone marrow function is defined as follows:

   Blood routine (no blood transfusion, no G-CSF, no medication correction within 14 days before screening) :

   Neutrophil count (ANC)≥1,500/mm3(1.5×109/L); Platelet count (PLT)≥100,000/mm3(100×109/L); Hemoglobin (Hb)≥9g/dL(90g/L);

   Blood biochemical:

   Serum creatinine (Cr)≤1.5× upper limit of normal (ULN) or creatinine clearance (Cockroft-Gault formula)≥60ml/min; Total bilirubin (TBIL)≤1.5×ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤2.5×ULN, and subjects with liver metastases should ≤5×ULN;

   Blood coagulation function:

   International normalized ratio (INR)≤1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT)≤1.5×ULN;
9. Urine routine: urinary protein <2+; If urine protein ≥2+, 24-hour urine protein quantification must show protein ≤1g;
10. Thyroid function: Thyroid stimulating hormone (TSH)≤ULN; FT3(T3) and FT4(T4) levels should be examined if they are abnormal, and normal FT3(T3) and FT4(T4) levels can be selected.
11. Female subjects of reproductive age must have a negative serum pregnancy test within 7 days prior to medication and be willing to use a medically approved highly effective contraceptive (e.g., intrauterine device, birth control pill, or condom) during the study period and within 3 months after the last administration of the study drug; Male subjects with a female partner of reproductive age were required to undergo surgical sterilization or consent to use an effective method of contraception during the study period and for 3 months after the last study dose.
12. I have AGREED and signed the informed CONSENT, and I am willing AND ABLE TO comply with the planned visit, study treatment, laboratory tests and other trial procedures.

Exclusion Criteria:

1. C1D1 received the following treatments in the previous 4 weeks:

   Radiotherapy, surgery, chemotherapy, immunotherapy for tumors. Other investigational drugs. Get live attenuated vaccine.
2. Surgery and/or radiation therapy for bone and soft tissue sarcomas were planned during the study.
3. Previous use of immunosuppressive drugs within 14 days prior to C1D1, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (i.e., no more than 10mg/ day of prednisolone or an equivalent physiological dose of another corticosteroid).
4. Severe infection (such as the need for intravenous antibiotic, antifungal, or antiviral medication) within 4 weeks prior to C1D1, or unexplained fever >38.5°C during the screening period/before the first dose.
5. Hypertension that is not well controlled with antihypertensive medication (systolic blood pressure > 140 mmHg or diastolic blood pressure >90mmHg).
6. Significant bleeding symptoms or clear bleeding tendency occurred within 3 months before C1D1, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, vasculitis, etc. Or arteriovenous thrombotic events occurring within 6 months before C1D1, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism; Long-term anticoagulant therapy with warfarin or heparin or long-term antiplatelet therapy (aspirin ≥300mg/ day or clopidogrel ≥75mg/ day) may be required.
7. Active heart disease in the 6 months prior to C1D1, including myocardial infarction and severe/unstable angina pectoris. Left ventricular ejection fraction <50% on echocardiography, poorly controlled arrhythmias (including QTcF interval >450ms in men and >470ms in women).
8. C1D1 had been diagnosed with any other malignancy within 3 years prior to C1D1, except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix.
9. Known allergy to the study drug or any of its excipients.
10. Human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B surface antigen positive and HBVDNA≥500IU/ml), and hepatitis C (hepatitis C antibody positive and HCV-RNA above the detection limit of the assay).
11. Concomitant diseases (e.g., poorly controlled hypertension, severe diabetes,neurological or mental disorders, etc.) or any other conditions that, in the judgment of the investigator, seriously endanger the safety of the subjects, may confounding the results of the study, or interfere with the completion of the study.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to approximately 24months
  From the start of treatment to the onset of disease progression or death of the patient
Objective response rate | Up to approximately 24months
  Until the tumor progresses or the patient dies or is lost to follow-up or cannot tolerate it

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No